CLINICAL TRIAL: NCT06314152
Title: A Comparative Study of 3-point With 1-point Mesh Fixation in TAPP for Inguinal Hernia
Brief Title: 3-point With 1-point Mesh Fixation in TAPP for Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Collaborators: Guang'an People's Hospital (Unknown); Pengan County People's Hospital (Other); People's Hospital of Yilong County (Unknown); Nanbu Hospital of County Chinese Medicine (Other); Langzhong People's Hospital (Unknown); Langzhong Traditional Chinese Medicine Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023032
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-11

CONDITIONS: Inguinal Hernia; Chronic Pain; Seroma; Recurrent; Infections; Hematoma
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain; Seroma; Recurrence; Infections; Hematoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3-point fixation group (Experimental): During laparoscopic transabdominal preperitoneal inguinal hernia repair, lightweight Mesh Fixation with 3-point Fixation. First fixation is in cooper ligament. Second fixation is in the back of rectus abdominis. Third fixation is in the later of tractus iliopubicus.
  Interventions: Procedure: Lightweight mesh fixation in 3 points or 1 point
- 1-point fixation group (Active Comparator): During laparoscopic transabdominal preperitoneal inguinal hernia repair, lightweight Mesh Fixation with 1-point Fixation in the back of rectus abdominis.
  Interventions: Procedure: Lightweight mesh fixation in 3 points or 1 point

INTERVENTIONS:
Procedure: Lightweight mesh fixation in 3 points or 1 point — Lightweight mesh fixation in 3 points

SUMMARY:
This study was designed to compare the outcome of 3 point with 1 point lightweight mesh fixation in TAPP surgery for patients with inguinal hernia. The main outcome include seroma, chronic pain, recurrence, et al.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral inguinal hernia according to preoperative physical examination and imaging examination.

The inclusion criteria were as follows: primary inguinal hernia.

Exclusion Criteria:

* Age below 18 years or older than 80. recurrent hernia, incarcerated hernia, strangulated hernia, and other types of hernias.

Patients not suitable for general anesthesia. Patients requiring open surgery; patients requiring emergency surgery Loss to follow-up or communication difficulties, or poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Rate of postoperative pain | 6 months
  The visual analog scale (VAS) was adopted for pain evaluation 2 days, 3 months, and 6 months postoperatively. The scale range from 0 to 10, with 0 meaning no pain and 10 meaning the worst pain.
Rate of recurrence | 1 month,3 months,6 months and 12 months after surgery
  Hernia recurrenceFollow up by physical examination, ultrasonography and telephone at 1 month,3 months,6 months and 12 months after surgery about the rate of hernia recurrence.

SECONDARY OUTCOMES:
Rate of postoperative complications | 6 months
  Including infection, seroma, hematoma

CONTACTS AND LOCATIONS:
Locations (1):
- Yunhong Tian, Nanchong, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided